CLINICAL TRIAL: NCT02802813
Title: A Randomised, Single-blinded Controlled Treatment Trial of Subclinical Vivax Infections With Primaquine in Nong Province, Laos
Brief Title: P.Vivax Treatment Trial
Acronym: Lao Pv
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LOMWRU1601
Record Dates: First submitted 2016-05-27; First posted 2016-06-16 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2017-08

CONDITIONS: Plasmodium Vivax
Keywords: Single-blinded controlled trial; Primaquine
MeSH Terms: conditions — Malaria, Vivax | interventions — Primaquine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention arm (Active Comparator): Dihydroartemisinin-piperaquine (DP) therapy plus 14 days of supervised primaquine (7mg/kg total dose) administered once per day (0.5 mg/kg).
  Interventions: Drug: Dihydroartemisinin-piperaquine (DP) + Primaquine (PQ)
- Control arm (Placebo Comparator): Dihydroartemisinin-piperaquine therapy plus 14 days identical placebo not containing primaquine.
  Interventions: Drug: Dihydroartemisinin-piperaquine (DP) + Primaquine (PQ) placebo

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine (DP) + Primaquine (PQ)
  Arms: Intervention arm
Drug: Dihydroartemisinin-piperaquine (DP) + Primaquine (PQ) placebo
  Arms: Control arm

SUMMARY:
This study aims to determine whether a 14 day course of 0.5 mg/kg/day primaquine can eliminate subclinical P. vivax infections detected by high volume ultra-sensitive PCR (uPCR).

DETAILED DESCRIPTION:
This is a randomized, Single blind trial in G6PD normal participants with subclinical P. vivax infections in Laos. Participants with subclinical P. vivax infections and those meeting the enrolment criteria will be randomly assigned to one of two treatment arms:

* Intervention: Dihydroartemisinin-piperaquine (DP) therapy 3 days dosing plus 14 days of supervised primaquine (7mg/kg total dose) administered once per day (0.5 mg/kg/day).
* Control arm: Dihydroartemisinin-piperaquine (DP) 3 days dosing therapy plus 14 days identical primaquine placebo.

Participants found to be G6PD deficient (G6PDd) will be treated with primaquine 0.75mg/kg/week for 8 weeks according to WHO recommendations. Primaquine and placebo will be administered with food (biscuits), which has been shown to reduce gastrointestinal side effects. All doses of study drugs will be supervised. If participants cannot visit the study centre, or fail to attend during the 14 days of supervised therapy, team members will visit them in their homes, schools or work to ensure complete dosing.

Findings:

The study showed that a 14-day course of primaquine added to mass drug administration with dihydroartemisinin-piperaquine prevented recurrent asymptomatic P. vivax infections (doi: 10.1186/s12936-019-3091-5)

ELIGIBILITY:
Inclusion Criteria:

* Participants with subclinical mono- or mixed P. vivax infections (uPCR) can be enrolled.
* Able to participate as decided by the investigators, and willing to comply with the study requirements and follow-up.
* A participant (or parent/guardian of children below age of consent) is willing and able to give written informed consent to participate in the trial.

Exclusion Criteria:

* Currently pregnant or breastfeeding (female of child-bearing age).
* Inability to tolerate oral treatment.
* Previous episode of haemolysis or severe haemoglobinuria following primaquine.
* Known hypersensitivity or allergy to the study drugs.
* Blood transfusion in last 90 days, since this can mask G6PD deficiency.
* An acute malaria episode requiring treatment.
* A febrile condition due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration).
* Anaemia (Haemoglobin (Hb) < 9 g/dL
* Presence of any condition which in the judgment of the investigator would place the participant at undue risk or interfere with the results of the study (e.g. serious underlying cardiac, renal or hepatic disease; severe malnutrition; HIV/AIDS; or severe febrile condition other than malaria); co-administration of other medication known to cause haemolysis or that could interfere with the assessment of antimalarial regimens.
* Currently taking medication known to interfere significantly with the pharmacokinetics of primaquine and the schizontocidal study drugs

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
The incidence rate of P. vivax parasitaemia in G6PD-normal participants | over 12 months
  the incidence rate will be detected by uPCR

SECONDARY OUTCOMES:
Time to P. vivax clearance | 12 months
  Detected by uPCR
The frequency of recurrent vivax infections (clinical and sub-clinical) | 12 months
The follow-up period required to detect a statistically significant difference in the frequency of recurrent subclinical P. vivax infections between treated and untreated participants | 12 months
  measured by uPCR
Number of participants with treatment related Adverse event. | 28 days
Number of participants with treatment related malaria episode | 12 months
Number of doses taken per participants | 14 days
Compare the percentage decrease in hemoglobin between those who receive primaquine and who those not receive primaquine | 12 months
Number of G6PD genotypes in participants with G6PD deficiency | 12 months
Number of P450 genotypes in participants with recurrent PV infection. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mayfong Mayxay, MD, Principal Investigator — Lao-Oxford-Mahosot Hospital Wellcome Trust Research Unit
Locations (1):
- Lao-Oxford-Mahosot Hospital-Wellcome Trust Research Unit, Vientiane, Laos

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Phommasone K, van Leth F, Imwong M, Henriques G, Pongvongsa T, Adhikari B, Peto TJ, Promnarate C, Dhorda M, Sirithiranont P, Mukaka M, Peerawaranun P, Day NPJ, Cobelens F, Dondorp AM, Newton PN, White NJ, von Seidlein L, Mayxay M. The use of ultrasensitive quantitative-PCR to assess the impact of primaquine on asymptomatic relapse of Plasmodium vivax infections: a randomized, controlled trial in Lao PDR. Malar J. 2020 Jan 3;19(1):4. doi: 10.1186/s12936-019-3091-5. PMID 31900172
- [Derived] von Seidlein L, Peerawaranun P, Mukaka M, Nosten FH, Nguyen TN, Hien TT, Tripura R, Peto TJ, Pongvongsa T, Phommasone K, Mayxay M, Imwong M, Watson J, Pukrittayakamee S, Day NPJ, Dondorp AM. The probability of a sequential Plasmodium vivax infection following asymptomatic Plasmodium falciparum and P. vivax infections in Myanmar, Vietnam, Cambodia, and Laos. Malar J. 2019 Dec 30;18(1):449. doi: 10.1186/s12936-019-3087-1. PMID 31888643